CLINICAL TRIAL: NCT05957718
Title: Effectiveness of TKTX Cream on Pain and Fear in Children During Venipuncture: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sherzad
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain; Fear of Pain; Venipuncture Site Numbness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TKTX Group (Experimental): In this group, We will use TKTX cream as a local anesthesia
  Interventions: Drug: TKTX cream
- Control Group (Placebo Comparator): In this group, we will use a Vasalin as Placebo
  Interventions: Drug: TKTX cream

INTERVENTIONS:
Drug: TKTX cream — TKTX cream was used in several studies on Tatto and laser
  Other Names: Placebo (Vasaline)

SUMMARY:
Venipuncture, the process of obtaining blood samples for diagnostic purposes, is a common medical procedure performed worldwide. However, it can be associated with varying levels of pain and discomfort for patients. Therefore, implementing effective pain management strategies during venipuncture is crucial to ensure patient comfort and improve the overall healthcare experience. This comprehensive overview aims to highlight the significance of pain management during venipuncture procedures.

This study will investigate the effects of a pharmacological approach on the pain that children experience during venipuncture in a randomized trial.

TKTX topical anesthetic cream is a new commercially available product. In this study, the cream will be used for a shorter period of time than other creams used in previous studies, and it will also be free of side effects as they have been in previous studies with other creams.

DETAILED DESCRIPTION:
Venipuncture is a common medical procedure involving the insertion of a needle into a vein, often causing discomfort and pain. To alleviate this pain, pharmacological approaches have been widely explored. The efficacy of these approaches in managing venipuncture-related pain is of utmost importance for both healthcare professionals and patients. Various pharmacological options have been studied, including topical anesthetics such as lidocaine creams or patches, local anesthetic injections like buffered lidocaine or ethyl chloride spray, and systemic analgesics such as nonsteroidal anti-inflammatory drugs (NSAIDs) or opioids.

You may experience some pain, often a brief sting, when the needle is inserted into and removed from your arm.

Non-pharmacological pain intervention is a prophylactic and complementary approach to reduce pain.

Ensuring safety and efficacy when performing blood draws on pediatric patients, while also accounting for their emotional and physical well-being is of utmost importance.

Pharmacological intervention: Topical anesthetics To reduce the discomfort generated by a venipuncture, the use of a topical anaesthetic cream is recommended prior to needle procedures, with options including EMLA (r), amethocaine and lidocaine.

Evaluating the effectiveness of these interventions requires considering factors like onset and duration of action, adequate pain relief achieved, patient satisfaction levels, and potential adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* School-age Children and
* Required needle procedures

Exclusion Criteria:

* Neurodevelopmental problems
* Chronic disease
* Taken Analgesic

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Scale Pain | 2-3 min. after procedure
  Was used to measure Children's pain scale

SECONDARY OUTCOMES:
Child Fear Scale | 2-3 min. after procedure
  Was used to measure Children's fear scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sherzad Khudeida Suleman, Duhok, Iraq

IPD SHARING:
Plan to Share IPD: No